CLINICAL TRIAL: NCT02376283
Title: Pharmacokinetics and Pharmacodynamics of Platelet P2Y12 Inhibitors in Patients Undergoing Percutaneous Coronary Intervention (PCI) for Acute Myocardial Infarction: A Pilot Study
Brief Title: P3AMI Antiplatelet Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-004-04-02-CARD
Record Dates: First submitted 2015-02-02; First posted 2015-03-03 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Heart Attack
Keywords: STEMI; NSTEMI; PPCI
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — Prasugrel Hydrochloride; Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- STEMI prasugrel (Other): Patients with diabetes mellitus admitted with STEMI who are under 75 years of age and greater than 60Kg in weight receiving Prasugrel Loading (60mg) and maintenance (10mg per day).
  Interventions: Drug: Prasugrel
- STEMI clopidogrel (Other): Patients admitted with STEMI over the age of 75 or under 60 Kg receiving clopidogrel loading (600 mg) and then maintenance (75mg per day).
  Interventions: Drug: Clopidogrel
- NSTEMI clopidogrel (Other): Patients admitted with NSTEMI/UA over the age of 75 or under 60 Kg receiving clopidogrel loading (600 mg) and then maintenance (75mg per day).
  Interventions: Drug: Clopidogrel
- Patients with NSTEMI (Other): who are under 75 years of age and greater than 60Kg in weight receiving Prasugrel loading (60mg) however: - i. After sample collection patients treated with intracoronary stent placement on the same day as loading will receive prasugrel maintenance dose (10mg per day) as per licensing agreement for prasugrel ii. After sample collection patients who are not stented after loading will receive clopidogrel maintenance dose (75mg per day).
  Interventions: Drug: Prasugrel; Drug: Clopidogrel
- Patients admitted with STEMI receiving ticagrelor loading (Other): Patients admitted with STEMI receiving ticagrelor loading (180 mg) and then maintenance (90mg bd per day)
  Interventions: Drug: ticagrelor
- Patients Admitted with NSTEMI receiving ticagrelor loading (Other): Patients Admitted with NSTEMI receiving ticagrelor loading (180 mg) and then maintenance (90mg bd per day).
  Interventions: Drug: ticagrelor

INTERVENTIONS:
Drug: Prasugrel
  Arms: Patients with NSTEMI; STEMI prasugrel
Drug: Clopidogrel
  Arms: NSTEMI clopidogrel; Patients with NSTEMI; STEMI clopidogrel
Drug: ticagrelor
  Arms: Patients Admitted with NSTEMI receiving ticagrelor loading; Patients admitted with STEMI receiving ticagrelor loading

SUMMARY:
Major heart attacks are caused by a numerous factors, including sudden clot formation in a coronary artery leading to a blockage and heart muscle death. The clots are largely made of sticky clotting blood cells (platelets). A patient having a major heart attack is treated with emergency primary percutaneous coronary intervention (PPCI) where a wire and balloon are used to reopen the coronary artery and a stent (a slotted metal tube) is placed to keep the artery open.

Aspirin, and one of two other antiplatelet drugs (prasugrel or ticagrelor) are given prior to PPCI to prevent further clots formation. Both antiplatelet drugs are taken in tablet form and in healthy stable patients these drugs take at least 30 min to 2 hours to exert an adequate effect. Often PPCI procedures are performed well within this timescale. It is possible that having a major heart attack limits the bodies ability to absorb the drugs also.

In this study, patients with major or minor heart attacks will be given either prasugrel or ticagrelor as per licensed indications and guideline recommendations. A 15 ml blood sample will be taken at first balloon inflation to reopen the blocked artery, then after 20 minutes, 60 minutes, and 4 hours after taking the drugs. Each blood sample will be subjected to a variety of tests to determine antiplatelet drug activity.

This study will identify which of the two agents used are working effectively during PPCI, given the very short timescales involved. It will also show if patients with major heart attacks absorb the drugs less well than patients with less severe heart attacks. In the future it might be that an intravenous agent will be more valuable in the setting of PPCI.

DETAILED DESCRIPTION:
This is a pilot study by design, which will be nonrandomized in nature. A total of 90 subjects will be included in the study distributed equally into 6 patient groups which have been carefully selected so that all patients will receive antiplatelet drugs as per current accepted NICE (National Institute for Health and aCare Excellence) guidelines and licensed indications.

In the current ethically approved protocol ver 1.4 (5/11/12) Groups 1,3 and 4 have already been recruited to and a full data set has been collected; Group 1 STEMI (ST-segment elevation myocardial infarction) prasugrel Group 3 STEMI clopidogrel Group 4 NSTEMI (Non-ST segment elevation myocardial infarction) clopidogrel

The current protocol allows for a specific group of NSTEMI patients (diabetic <75 years of age, >60 kg) treated with prasugrel to be recruited. The restrictive nature of these criteria would not allow us to make a direct comparison to STEMI patients treated with prasugrel. In light of this the eligibility criteria has been widened for NSTEMI patients to be treated with prasugrel. The proposed NSTEMI criteria is as follows:

1. Group 2: Patients with NSTEMI who are under 75 years of age and greater than 60kg in weight receive prasugrel loading (60mg) (in line with the manufacturers recommendations and licensing) after the 4 hour sample collection period those patients who are treated with percutaneous coronary intervention will receive prasugrel at a maintenance dose of 10mg daily (in line with NICE recommendations and local guidelines), those patients who do not proceed to be treated with percutaneous coronary intervention will be switched to clopidogrel 75mg daily (in line with NICE recommendations and local guidelines) on the following day.

   The investigators also propose to include recruitment of the following two groups in which ticagrelor will prescribed in accordance with NICE guidance and licenced indications:
2. Group 5: Patients admitted with STEMI receiving ticagrelor loading (180 mg) and then maintenance (90mg bd per day)(in line with manufacturer's recommendations and licensing).
3. Group 6: Patients Admitted with NSTEMI receiving ticagrelor loading (180 mg) and then maintenance (90mg bd per day)(in line with manufacturer's recommendations and licensing) The investigators will only begin recruitment to groups 5 and 6 once patient recruitment is completed in group 2

PROCEDURE LOG:

STEMI patients will be identified following admission for PPCI. Patient consent for this group shall be a 2 stage process. Initially, a shortened patient information sheet shall be read to the patient on admission prior to PPCI as to not delay treatment. Once verbal consent has been obtained a P2Y12 inhibitor ticagrelor will be administered to the patient as per current local and national guidance. The time of loading dose will be carefully recorded and the patient transferred to the cardiac catheterization suite for PPCI. After the insertion of the radial or femoral sheath, 15 ml (approx 3 teaspoonfuls in volume) of whole blood will be drawn from this sheath at 20 minutes post dosing (or as close to this time point as practicable) and also at the first balloon inflation time. A further 15 ml will be taken at 60 minutes post dosing (or as close as is practicable). The second stage of consent will occur after PPCI when the patient has been transferred to the ward and is pain free and has been able to rest. At this stage a full patient information sheet shall be given to the patient to read and written consent will be sought. A final 15ml blood sample will be taken after 4 hours post dosing, after which the patient's participation in this study will come to an end.

NSTEMI/UA (Unstable Angina) Potential patients will be approached by a member of the research team, who will offer the patient a full written patient information sheet and obtain written consent. Following consent the patient will have been administered a P2Y12 inhibitor (prasugrel or ticagrelor). The time of loading dose will be carefully recorded. 15 ml (approx 3 teaspoonfuls in volume ) of blood will be taken at 20 minutes, 60 minutes and then 4 hours post dosing, after which the patient's participation in this study will come to an end.

For both STEMI and NSTEMI/UA groups, aspirin will already have been given in the ambulance and will be assessed at 20 minutes after P2Y12 inhibitor loading and again at 60 minutes.

Each blood sample taken will undergo a series of tests which will encompass the presence and function of the antiplatelet medication after a patient has suffered either a major or minor heart attack.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with STEMI for PCI (characterized by chest discomfort, and prominent STsegment elevation)
2. Patients presenting with NSTEMI (characterized by chest discomfort, raised levels of myocardial enzymes and/or STsegment depression or prominent T wave inversion)
3. Able to give verbal consent (STEMI patients pre procedure) and/or written consent (STEMI after procedure and NSTEMI patients prior to enrolment).
4. Age>18 years of age
5. Able to take Aspirin and either prasugrel or ticagrelor.
6. Have no concurrent septic or inflammatory illness
7. Thienopyridine naive

Exclusion Criteria:

1. Be unable to provide verbal and written consent
2. Allergic to aspirin or any of the P2Y12 antagonists in the trial
3. Have preexisting cardiogenic shock
4. Have a concurrent septic or inflammatory disease e.g. rheumatoid arthritis, lupus, pneumonia.
5. Already taking a P2Y12 inhibitor
6. Known bleeding diathesis
7. Patients under 75 years of age or under 60 kg or those who have had a previous stroke/transient ischaemic attack, will not be eligible for prasugrel but rather ticagrelor.
8. Patients with a history of intracranial haemorrhage will not receive prasugrel or ticagrelor but rather will receive treatment with clopidogrel.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Cotton, MD, FRCP, Study Director — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Clopidogrel: STEMI (ST-segment elevation myocardial infarction) (n = 14) and NSTEMI (Non-ST segment elevation myocardial infarction) (n = 13) patients were administered a clopidogrel 600mg loading dose and whole blood samples (15ml) for pharmacodynamic assessment of the degree of platelet inhibition were obtained. Plasma samples to allow for pharmacokinetic quantification of active metabolites were extracted from whole blood samples collected. Samples were collected at 20 minutes, 60 minutes and 240 minutes post loading. In the STEMI group an additional sample was collected at the time of angioplasty.
  The participants involvement in the study ceased following the collection of the 240-minute blood sample.
- Prasugrel: STEMI (n = 15) and NSTEMI (n = 15) patients were administered a prasugrel 90mg loading dose and whole blood samples (15ml) for pharmacodynamic assessment of the degree of platelet inhibition were obtained. Plasma samples to allow for pharmacokinetic quantification of active metabolites were extracted from whole blood samples collected. Samples were collected at 20 minutes, 60 minutes and 240 minutes post loading. In the STEMI group an additional sample was collected at the time of angioplasty.
  The participants involvement in the study ceased following the collection of the 240-minute blood sample.
- Ticagrelor: STEMI (n = 15) and NSTEMI (n = 15) patients were administered a ticagrelor 180mg loading dose and whole blood samples (15ml) for pharmacodynamic assessment of the degree of platelet inhibition and pharmacokinetic quantification of parent compound and active metabolites were collected. Samples were collected at 20 minutes, 60 minutes and 240 minutes post loading. In the STEMI group an additional sample was collected at the time of angioplasty.
  The participants involvement in the study ceased following the collection of the 240-minute blood sample.
Period: Overall Study
Arm/Group | Clopidogrel | Prasugrel | Ticagrelor
Started | 27 | 30 | 30
Completed | 27 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clopidogrel: STEMI (n = 14) and NSTEMI (n = 13) patients were administered a clopidogrel 600mg loading dose and whole blood samples (15ml) for pharmacodynamic assessment of the degree of platelet inhibition were obtained. Plasma samples to allow for pharmacokinetic quantification of active metabolites were extracted from whole blood samples collected. Samples were collected at 20 minutes, 60 minutes and 240 minutes post loading. In the STEMI group an additional sample was collected at the time of angioplasty.
  The participants involvement in the study ceased following the collection of the 240-minute blood sample.
- Total: Total of all reporting groups
Arm/Group | Clopidogrel | Prasugrel | Ticagrelor | Total
Number analyzed (Participants) | 27 | 30 | 30 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 19 | 13 | 41
  >=65 years | 18 | 11 | 17 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 6 | 19
  Male | 19 | 25 | 24 | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 27 | 30 | 30 | 87

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamic Assessment of Degree of Platelet Inhibition as Determined by Verify Now Point of Care Assay and Expressed as P2Y12 Reaction Units (PRU)
Time Frame: Balloon Inflation as Baseline, 20, 60, 240 minutes
Population: The overall group consists of STEMI and NSTEMI participants -outcome measure is broken down into the time points for each specific sub-group reported separately by Row. These two categories represent a subpopulation within the Overall Number of Participants Analyzed, therefore it has been indicated how many participants were analyzed for each Row.
Measure: Mean (Standard Deviation); unit: P2Y12 reaction units (PRU)
Arm/Group | Clopidogrel | Prasugrel | Ticagrelor
Number analyzed (Participants) | 27 | 30 | 30
P2Y12 reaction units (PRU)
  STEMI at 20 mins: number analyzed (Participants) | 14 | 15 | 15
  STEMI at 20 mins | 270.23 (38.56) | 247.73 (48.78) | 256.73 (50.81)
  STEMI at balloon inflation: number analyzed (Participants) | 14 | 15 | 15
  STEMI at balloon inflation | 286.46 (33.12) | 253.73 (57.17) | 257.93 (61.12)
  STEMI at 60 mins: number analyzed (Participants) | 14 | 15 | 15
  STEMI at 60 mins | 293.46 (31.68) | 262.87 (43.43) | 225.20 (82.70)
  STEMI at 240 mins: number analyzed (Participants) | 14 | 15 | 15
  STEMI at 240 mins | 226.42 (69.44) | 128.64 (89.16) | 176.27 (84.92)
  NSTEMI at 20 mins: number analyzed (Participants) | 13 | 15 | 15
  NSTEMI at 20 mins | 213.21 (51.74) | 125.80 (89.34) | 172.80 (92.54)
  NSTEMI at 60 mins: number analyzed (Participants) | 13 | 15 | 15
  NSTEMI at 60 mins | 227.36 (61.19) | 76.93 (99.24) | 114.20 (122.22)
  NSTEMI at 240 mins: number analyzed (Participants) | 13 | 15 | 15
  NSTEMI at 240 mins | 214.00 (69.98) | 31.87 (45.52) | 23.00 (18.94)
Statistical Analysis 1: Comparison: Clopidogrel vs Prasugrel vs Ticagrelor; Continuous variables expressed as mean ± SD (standard deviation) and categorical variables as frequencies (%).Continuous variables analysed individually using student's independent sample t-tests. Categorical variables assessed using separate Fisher's exact (Chi-square) test; Test type: Other — A p value < 0.05 was considered to be statistically significant.Comparison of means between groups assessed using ANOVA allowing comparison of more than 2 means and enabled assessment made of the relationship between different drugs (clopidogrel vs prasugrel vs ticagrelor), different clinical states (STEMI vs NSTEMI/UA (Unstable angina)) and different time points; p < 0.05, ANOVA — Assessment made of relationship between groups-clop vs pras vs tic,rows of STEMI vs NSTEMI/UA and different time points.P-values reported are calculated values based on data collated during sample collection and review of clinical characteristics
Statistical Analysis 2: Comparison: Clopidogrel vs Prasugrel vs Ticagrelor; STEMI- clop vs prasl vs tic; Test type: Other — Comparison of means between groups assessed using ANOVA allowing comparison of more than 2 means and enabled assessment made of the relationship between different drugs (clopidogrel vs prasugrel vs ticagrelor), different clinical states (STEMI vs NSTEMI/UA (Unstable angina)) and different time points; p < 0.0001, ANOVA; ANOVA F(3,36) = 12.282
Statistical Analysis 3: Comparison: Clopidogrel vs Prasugrel vs Ticagrelor; NSTEMI- clopidogrel vs prasugrel vs ticagrelor; Test type: Other — [test comment as in outcome 1, analysis 2]; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; ANOVA F(2,40) = 29.097

2. Primary Outcome: Pharmacokinetic Quantification of Plasma Concentration of Clopidogrel and Prasugrel Active Metabolite and Ticagrelor Parent Compound and Active Metabolite Assessed Using Liquid Chromatography in Tandem With Mass Spectrometry (LC-MS/MS) Expressed as ng/ml
Description: The parent compound of Ticagrelor was also analysed within the same patient group of Ticagrelor as it is a directly acting agent that does not require metabolic conversion to its active form.
Time Frame: Balloon Inflation as Baseline, 20, 60, 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/ml
Groups:
- Ticagrelor Parent Compound: STEMI/NSTEMI patients. (Ticagrelor was used in our centre only after the use of prasugrel was discontinued) The parent compound was also analysed as it is a directly acting agent that does not require metabolic conversion to its active form
Arm/Group | Clopidogrel | Prasugrel | Ticagrelor | Ticagrelor Parent Compound
Number analyzed (Participants) | 27 | 30 | 30 | 30
ng/ml
  STEMI at 20 mins: number analyzed (Participants) | 14 | 15 | 15 | 15
  STEMI at 20 mins | 39.12 (16.17) | 14.27 (8.80) | 0.16 (0.16) | 9.04 (4.12)
  STEMI at balloon inflation: number analyzed (Participants) | 14 | 15 | 15 | 15
  STEMI at balloon inflation | 107.83 (44.08) | 24.20 (13.07) | 1.64 (1.17) | 28.56 (12.58)
  STEMI at 60 mins: number analyzed (Participants) | 14 | 15 | 15 | 15
  STEMI at 60 mins | 71.02 (27.21) | 36.86 (13.27) | 14.43 (7.28) | 47.13 (24.09)
  STEMI at 240 mins: number analyzed (Participants) | 14 | 15 | 15 | 15
  STEMI at 240 mins | 32.41 (6.71) | 38.44 (7.59) | 53.38 (25.21) | 84.92 (42.00)
  NSTEMI at 20 mins: number analyzed (Participants) | 13 | 15 | 15 | 15
  NSTEMI at 20 mins | 41.99 (25.27) | 515.80 (126.84) | 7.72 (5.10) | 22.78 (10.27)
  NSTEMI at 60 mins: number analyzed (Participants) | 13 | 15 | 15 | 15
  NSTEMI at 60 mins | 93.35 (49.65) | 194.59 (29.97) | 58.40 (25.41) | 84.13 (34.02)
  NSTEMI at 240 mins: number analyzed (Participants) | 13 | 15 | 15 | 15
  NSTEMI at 240 mins | 27.71 (6.90) | 36.80 (4.59) | 113.59 (19.20) | 140.61 (36.31)
Statistical Analysis 1: Comparison: Clopidogrel vs Prasugrel vs Ticagrelor vs Ticagrelor Parent Compound; Continuous variables were expressed as mean ± SEM (Standard Error of Measurement) and categorical variables as frequencies (%). Continuous variables were analysed individually using student's independent sample t-tests. Categorical variables were assessed using separate Fisher's exact (Chi-square) test; Test type: Other — Comparison of means between groups was assessed using analysis of variance (ANOVA) technique. ANOVA allowed for a comparison of more than two means and enabled an assessment to be made of the relationship between, different drugs (clopidogrel active metabolite vs prasugrel active metabolite vs ticagrelor parent compound and active metabolite), different clinical states (STEMI vs NSTEMI/UA (Unstable angina)) and different time points; p < 0.05, ANOVA — Assessment made of relationship between groups-clop vs pras vs tic, rows of STEMI vs NSTEMI/UA and different time points. P-values reported are calculated values based on data collated during sample collection and review of clinical characteristics
Statistical Analysis 2: Comparison: Clopidogrel vs Prasugrel vs Ticagrelor vs Ticagrelor Parent Compound; STEMI- different drugs (as stated above); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.123, ANOVA; ANOVA F(6,56)=1.707
Statistical Analysis 3: Comparison: Clopidogrel vs Prasugrel vs Ticagrelor vs Ticagrelor Parent Compound; NSTEMI- different drugs (as stated above); Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; ANOVA F(4,62)=18.932

3. Secondary Outcome: Pharmacodynamic Assessment of Degree of Platelet Inhibition as Determined by VASP (Vasodilator Stimulated Phosphoprotein Phosphorylation) Flow Cytometry and Expressed as %PRI (Platelet Reactivity Index)
Time Frame: Balloon Inflation as Baseline, 20, 60, 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: %PRI
Arm/Group | Clopidogrel | Prasugrel | Ticagrelor
Number analyzed (Participants) | 27 | 30 | 30
%PRI
  STEMI at 20 mins: number analyzed (Participants) | 14 | 15 | 15
  STEMI at 20 mins | 76.29 (8.77) | 46.25 (13.91) | 79.75 (9.20)
  STEMI at balloon inflation: number analyzed (Participants) | 14 | 15 | 15
  STEMI at balloon inflation | 74.86 (9.00) | 41.13 (12.71) | 74.63 (11.42)
  STEMI at 60 mins: number analyzed (Participants) | 14 | 15 | 15
  STEMI at 60 mins | 71.57 (11.68) | 50.50 (11.88) | 76.25 (11.12)
  STEMI at 240 mins: number analyzed (Participants) | 14 | 15 | 15
  STEMI at 240 mins | 63.14 (13.26) | 57.00 (10.39) | 51.38 (14.06)
  NSTEMI at 20 mins: number analyzed (Participants) | 13 | 15 | 15
  NSTEMI at 20 mins | 75.17 (2.74) | 33.27 (10.66) | 62.00 (8.79)
  NSTEMI at 60 mins: number analyzed (Participants) | 13 | 15 | 15
  NSTEMI at 60 mins | 76.75 (4.35) | 21.91 (9.72) | 33.17 (17.73)
  NSTEMI at 240 mins: number analyzed (Participants) | 13 | 15 | 15
  NSTEMI at 240 mins | 61.83 (5.82) | 15.18 (5.85) | 20.17 (10.48)
Statistical Analysis 1: Comparison: Clopidogrel vs Prasugrel vs Ticagrelor; Continuous variables were expressed as mean ± SD and categorical variables as frequencies (%). Continuous variables were analysed individually using student's independent sample t-tests. Categorical variables were assessed using separate Fisher's exact (Chi-square) test; Test type: Other — Comparison of means between groups was assessed using analysis of variance (ANOVA) technique. ANOVA allowed for a comparison of more than two means and enabled an assessment to be made of the relationship between, different drugs (clopidogrel vs prasugrel vs ticagrelor), different clinical states (STEMI vs NSTEMI/UA) and different time points; p < 0.05, ANOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Clopidogrel vs Prasugrel vs Ticagrelor; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.810, ANOVA — STEMI- clopidogrel vs prasugrel vs ticagrelor; ANOVA F(3,17) = 0.321
Statistical Analysis 3: Comparison: Clopidogrel vs Ticagrelor; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p < 0.0001, ANOVA — NSTEMI- clopi vs pras vs tic; ANOVA F(2,25) = 14.103

ADVERSE EVENTS:
Time Frame: 4 hours
Arm/Group | Clopidogrel | Prasugrel | Ticagrelor
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/27 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT02376283/Prot_SAP_000.pdf